CLINICAL TRIAL: NCT00493571
Title: Phase I Study of Gimatecan in Patients With Myelodysplastic Syndromes
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Novartis (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2006-0943; NCI-2010-00622 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2007-06-27; First posted 2007-06-28 (Estimated); Last update posted 2015-05-13 (Estimated); Status verified 2015-05

CONDITIONS: Myelodysplastic Syndromes; MDS
Keywords: Myelodysplastic Syndromes; MDS; Gimatecan; Leukemia
MeSH Terms: conditions — Myelodysplastic Syndromes; Leukemia | interventions — ST 1481

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Gimatecan (Experimental): Gimatecan Starting dose: 0.6 mg capsules administered orally once daily.
  Interventions: Drug: Gimatecan

INTERVENTIONS:
Drug: Gimatecan — Starting dose: 0.6 mg capsules administered orally once daily.

SUMMARY:
The goal of this clinical research study is to find the highest tolerable dose of gimatecan that can be given to treat myelodysplastic syndrome (MDS).

DETAILED DESCRIPTION:
The Study Drug:

Gimatecan is designed to block the function of an important protein (topoisomerase I) in cancer cells that helps repair damage to DNA (the genetic material of cells). When this protein is blocked, cancer cells may die.

Screening Tests:

Before you can start receiving the study drug, you will have what are called "screening tests." These tests will help the doctor decide if you are eligible to take part in this study.

* You will have a physical exam.
* Your complete medical history will be recorded.
* Your vital signs (blood pressure, pulse, breathing rate, and temperature), height, and weight will be measured.
* You will be asked how well you are able to perform the normal activities of daily living (a performance status evaluation).
* You will be asked about any medications you may be taking.
* Blood (about 1 tablespoon) will be drawn for routine tests.
* Women who are able to have children must have a negative blood (about 2 teaspoons) or urine pregnancy test.
* You will have a bone marrow aspirate performed. To collect a bone marrow aspirate, an area of the hip is numbed with anesthetic, and a small amount of bone marrow is withdrawn through a large needle.
* If your doctor thinks it is necessary, you will have a bone marrow biopsy when you have the bone marrow aspirate done. To collect a bone marrow biopsy, an area of the hip is numbed with anesthetic, and a small amount of bone marrow and bone is withdrawn through a large needle.
* You will complete a questionnaire to see how the disease may be affecting your ability to do your daily activities. The questionnaire will take about 15 minutes to complete.

Study Drug Dose Level:

If you are found to be eligible to take part in this study, the amount of study drug you receive will be based on when you join the study. Three (3) to 6 participants will be enrolled in this study and given a certain dose. If they do not experience intolerable side effects, the next 3-6 participants enrolled will receive a higher dose. This process will continue until researchers find the highest dose of the drug that can be given without causing serious or intolerable side effects. The study doctor will tell you what dose you will be receiving and how this compares to the doses other participants have received.

Study Drug Administration:

You will take gimatecan on Days 1-5. On Days 6-28, you will take no study drug. Each 28-day period is called a study "cycle." If your doctor thinks it is necessary, your study cycles may be shortened so that you will receive the study drug more often.

You will take the medication on an empty stomach, swallowing the capsules whole. You should not eat for 1 hour after taking the medication. If you take other medications while you are on this study, they must be taken 4 hours before or after you take gimatecan.

Study Visits:

Blood (about 2 tablespoons each time) will be drawn for routine tests every 1-4 weeks for the length of this study. Most of these blood tests will be done once a week, but some will only be done once every 4 weeks.

You will have a physical exam every 4 weeks for the first 3 months, then every 3 months.

At the end of Cycle 1, and then every 9-12 weeks after that, you will have a bone marrow aspirate and/or biopsy. Bone marrow biopsies and aspirates may be collected more often if your study doctor thinks it is necessary.

Once per week for the first 3 cycles, you will complete a symptom questionnaire. This will be done either at a study visit, or you will be called by a member of study staff. The questionnaire will take about 15 minutes to complete.

Length of Study:

You can remain on this study for up to 12 months. If, after this time, it is considered that gimatecan is helping you, the study doctor will discuss the possibility of continuing the study drug therapy outside of this study. You may be taken off this study early if the disease gets worse or intolerable side effects occur.

End-of-Study Visit:

Once you are off this study, you will have an end-of-study visit, and the following tests will be performed.

* You will have a physical exam.
* You will be asked about any side effects you may be experiencing.
* Blood (about 4 teaspoons) will be drawn for routine tests.
* You will repeat the symptom questionnaire.

This is an investigational study. Gimatecan is not FDA approved or commercially available. It has been authorized for use in research only. Up to 30 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with MDS with >/= 5% blasts or IPSS risk group intermediate (1 or 2) or high (i.e., IPSS score 0.5 or higher).
2. Patients must have failed prior therapy with either chemotherapy (e.g., ara-C-based chemotherapy, etc) or biologic agents (e.g., hypomethylating agents, arsenic, thalidomide, CC5013, farnesyl transferase inhibitors, ATG, cyclosporine, etc).
3. Age >/= 18 years. Because no dosing or adverse event data are currently available on the use of Gimatecan in patients <18 years of age, children are excluded from this study but will be eligible for future pediatric single-agent trials, if applicable.
4. Eastern Cooperative Oncology Group (ECOG) performance status 0-2.
5. Patients must have normal organ function as defined below: 1) Total bilirubin: </= 1.5 x institutional upper limit of normal; 2) ALT(SGPT): </= 2.5 x institutional upper limit of normal; 3) Creatinine: </= 1.5 x institutional upper limit of normal.
6. The effects of Gimatecan on the developing human fetus at the recommended therapeutic dose are unknown. For this reason women of child-bearing potential (ie, not post-menopausal for at least 12 months and not surgically sterile) and men must agree to use double-barrier contraception prior to study entry, for the duration of study participation, and for 3 months following discontinuation of study treatment. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately.
7. Ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria:

1. Patients who have received only supportive care (transfusions and/or hematopoietic growth factors) for MDS.
2. Patients who have had chemotherapy or radiotherapy within 4 weeks or 5 half-lives of the agent in question (6 weeks for nitrosoureas or mitomycin C), whichever is greater, prior to entering the study or those who have not recovered to at least grade 1 from adverse events due to agents administered more than 4 weeks earlier. The use of hydroxyurea is allowed up to 48 hours prior to the start of therapy with Gimatecan.
3. Uncontrolled intercurrent illness including, but not limited to, active uncontrolled infection, symptomatic congestive heart failure, unstable angina pectoris, symptomatic cardiac arrhythmia requiring and not responding to medical intervention, or psychiatric illness/social situations that would limit compliance with study requirements.
4. Women who are pregnant or breast-feeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2007-08; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of Gimatecan | Evaulate with each 28 Day Cycle
  For purposes of estimating the MTD, 5 dose levels of Gimatecan initially considered. These dose levels are 3 mg, 5 mg, 7.5 mg, 8.75 mg, and 10 mg orally per cycle. Dose escalation based on toxicities observed through the first cycle.

SECONDARY OUTCOMES:
Efficacy in terms of complete remission , complete remission w/ incomplete platelet or neutrophil recovery (CRp and CRn, respectively), partial remission , and hematologic improvement. | Up to 12 Months on Study
  Response criteria according to the International Working Group (Blood 2006; 108: 419-425). Responders are patients who obtain a Complete Response (CR), CRi, Partial Response (PR), with or without cytogenetic response, hematologic improvements, and morphologic leukemia-free state.

CONTACTS AND LOCATIONS:
Overall Officials: Jorge E. Cortes, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- The University of Texas M.D. Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: M.D. Anderson's website — http://mdanderson.org